CLINICAL TRIAL: NCT07091942
Title: Curative Therapy After Atezolizumab and Bevacizumab Treatment for Unresectable Hepatocellular Carcinoma: A Multinational Retrospective Study
Brief Title: Curative Therapy After Atezolizumab and Bevacizumab Treatment for Unresectable Hepatocellular Carcinoma
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government); Chi Mei Medical Hospital (Other); National Taiwan University Hospital Hsin-Chu Branch (Other); National Taiwan University (Other); Taichung Veterans General Hospital (Other); E-DA Hospital (Other); Chiayi Christian Hospital (Other); Srinagarind Hospital, Khon Kaen University (Other)
Responsible Party: Sponsor
Other Study IDs: 202504033RIPE
Record Dates: First submitted 2025-07-17; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Curative LRT cohort: Patients who received curative locoregional therapy after obtaining partial response after atezolizumab-bevacizumab treatment
- Comparative cohort: Patients who obtained completed or partial response after atezolizumab-bevacizumab treatment and did not receive curative locoregional therapy

SUMMARY:
Combination immunotherapy is currently the standard first-line systemic treatment for unresectable hepatocellular carcinoma (HCC). Approximately 30 % of patients treated with atezolizumab plus bevacizumab (Atezo-Bev) achieve complete or partial tumor response. Some patients who reach a partial response experience enough tumor regression to undergo curative therapies and subsequently attain a disease-free state. However, whether the prognosis of patients who become disease-free after curative therapy equals that of patients who achieve complete response with Atezo-Bev alone is unclear. Likewise, it remains uncertain whether patients who achieve partial response with Atezo-Bev and later undergo curative therapy fare better than those who remain in partial response without further curative treatment. Therefore, we designed this multinational, multicenter, retrospective chart-review study to address these questions.

Planned Cohorts

* Curative-therapy cohort: Patients with unresectable HCC who achieve partial response to Atezo-Bev and subsequently receive curative therapy-surgical resection, radiofrequency ablation, or definitive radiotherapy-to achieve a disease-free state.
* Control cohort: Patients with unresectable HCC who achieve complete or partial response to Atezo-Bev but do not undergo subsequent curative therapy.

Methods and End-points Data will be collected from no more than 30 hospitals worldwide, targeting roughly 400 patients in the curative-therapy cohort and 1,200 patients in the control cohort. Medical-record review will gather baseline characteristics, disease status, liver function, Atezo-Bev treatment details, curative-therapy specifics, treatment responses, and survival outcomes. The primary objective is to compare recurrence-free survival between the two cohorts. This retrospective study will close data collection on 31 March 2025.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or clinically (the presence of liver cirrhosis and typical HCC imaging findings by multi-phase CT or MRI) diagnosed HCC.
2. Received Atezo-Bev containing treatment as first-line systemic therapy for HCC
3. Patients with or without macrovascular invasion and main portal vein invasion before Atezo-Bev containing treatment can be enrolled
4. Patients with or without extrahepatic spread before Atezo-Bev containing treatment can be enrolled
5. Obtained CR or PR, according to RECIST version 1.1, to Atezo-Bev treatment

Exclusion Criteria:

1. Fibrolamellar carcinoma or mixed hepatocellular cholangiocarcinoma.
2. Received anti-CTLA4 antibodies simultaneously with Atezo-Bev Patients who received Atezo-Bev in combination with investigational drugs such as tiragolumab, relatlimab, and tocilizumab were allowed to enter the study.
3. Received locoregional therapy simultaneously with Atezo-Bev treatment, such as transarterial chemoembolization (TACE), hepatic arterial infusion of chemotherapy (HAIC), transarterial radioembolization, radiofrequency ablation, and microwave ablation before obtaining PR or not for curative intent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who obtained CR or PR, according to RECIST version 1.1, after receiving Atezo-Bev as first-line systemic therapy for clinically or histologically diagnosed HCC
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | From initiation of atezolizumab-bevacizumab treatment to disease recurrence or date of death from any cause, whichever came first, assessed up to 8 years

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Select, Taiwan